CLINICAL TRIAL: NCT02932358
Title: Effectiveness and Safety of a Flexible Family Visitation Model for Delirium Prevention in Adult Intensive Care Units: a Cluster-randomized, Crossover Trial
Brief Title: Effectiveness and Safety of a Flexible Family Visitation Model for Delirium Prevention in Adult Intensive Care Units: a Cluster-randomized, Crossover Trial (The ICU Visits Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Moinhos de Vento (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ICU Visits
Record Dates: First submitted 2016-10-11; First posted 2016-10-13 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Delirium
Keywords: Intensive care units; Delirium; Cross infection; Mortality; Length of stay; Burnout, Professional; Depression; Anxiety
MeSH Terms: conditions — Delirium; Cross Infection; Burnout, Professional; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The following interventions will be evaluated in the present study: restrictive family visitation model (intermittent visits according to local ICU regulation) and flexible family visitation model (12 consecutive hours per day). The unit of of concealed randomization is the ICU to minimize the risk of contamination, given that we intend to apply the intervention to the whole ICU multidisciplinary team. We will randomize ICUs to either an RFVM or to an FFVM as the initial intervention (T1). After enrollment of 25 ICU patients, there will be a 30-day period without recruitment to avoid contamination bias. After this period, each ICU will be assigned to an intervention contrary to that which initially receive (T2) until the enrollment of more 25 ICU patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexible Family Visitation Model (FFVM) (Active Comparator): In the FFVM, two or fewer family members will be allowed to visit the patient for up to 12 consecutive hours each day. In addition to family visitation, patients will be allowed to receive social visits in specific time intervals (according local ICU regulation). To have access to the FFVM, family members of ICU patients will have to attend a structured meeting at ICU in which they will receive orientations about the ICU environment, common ICU treatments, rehabilitation and basic infection control practices, multidisciplinary work at ICU and palliative treatment. Social visitors will not be required to attend the structured meeting.
  Interventions: Other: Flexible Family Visitation Model (FFVM)
- Restrictive Family Visitation Model (RFVM) (Active Comparator): In the RFVM, patients will be allowed to receive restricted visits according routine ICU practices, but respecting the maximum limit of 4.5 hours of visitation per day. Visitors will not be required to attend the structured meeting. The length of ICU visits will be similar to those of social visits in the FFVM.
  Interventions: Other: Restrictive Family Visitation Model (RFVM)

INTERVENTIONS:
Other: Flexible Family Visitation Model (FFVM) — Visitation to ICU patients allowed during the period of 12 consecutive hours per day.
  Arms: Flexible Family Visitation Model (FFVM)
Other: Restrictive Family Visitation Model (RFVM) — Visitation to ICU patients allowed during intermittent periods according local ICU regulation.
  Arms: Restrictive Family Visitation Model (RFVM)

SUMMARY:
A cluster-randomized crossover trial involving adult ICU patients, family members, and ICU professionals will be conducted. Forty medical-surgical Brazilian ICUs with visiting hours <4.5 h/day will be randomly assigned to either a restrictive family visitation model (RFVM) (visits according to local policies) or a flexible family visitation model (FFVM) (visitation during 12 consecutive hours per day) at a 1:1 ratio. After enrollment and follow-up of 25 patients, each ICU will be switched over to the other visitation model, until 25 more patients per site are enrolled and followed. The primary outcome will be the cumulative incidence of delirium among ICU patients, measured twice a day using the Confusion Assessment Method for the ICU. Secondary outcome measures will include daily hazard of delirium, ventilator-free days at day 7, any ICU-acquired infections, ICU length of stay, and all-cause hospital mortality among the patients; symptoms of anxiety and depression and satisfaction among the family members; and prevalence of symptoms of burnout among the ICU professionals. Tertiary outcomes will include need for antipsychotic agents and/or mechanical restraints, coma-free days at day 7, unplanned loss of invasive devices, and ICU-acquired pneumonia, urinary tract infection, or bloodstream infection among the patients; self-perception of involvement in patient care among the family members; and satisfaction among the ICU professionals.

ELIGIBILITY:
Inclusion Criteria:

* For ICUs: medical-surgical ICUs of of public and philanthropic Brazilian hospitals with restricted visitation policies(<4.5 hours/day).
* For Patients: Age ≥ 18 years, admission to the intensive care unit.
* For Patient's Family Members: nearest relative of the ICU patient recruited in the study and consent to participate in the study.
* For ICU Workers: ICU workers that assist patients in the ICU during the daytime for at least 20 hours per week and consent to participate in the study.

Exclusion Criteria:

* For ICUs: ICUs with structural or organizational impediments to extended visitation.
* For Patients: Subjects with coma (Richmond Agitation Sedation Scale -4 or -5) lasting > 96 hours from the moment of first evaluation for recruitment, or delirium at the baseline (positive Confusion Assessment Method for ICU) will be excluded. Individuals with cerebral death, aphasia, severe hearing deficit, a prediction of ICU length of stay < 48 hours, exclusively palliative treatment, or without a familiar member able to participate in extended ICU visits and those who are prisioners, unlikely to survive >24hs, re-admitted to the ICU after enrolment in the study will also be excluded.
* For Patient's Family Members: Another ICU patient's relative enrolled in the study; family members who don't speak Portuguese; Difficulty to answer the self-administered questionnaires (e.g.: illiteracy)
* For ICU Workers: ICU workers who have a prediction of withdrawal of ICU care activities >15 days during the study will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1650 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

PRIMARY OUTCOMES:
Incidence of Delirium among ICU patients | During ICU stay (from enrollment until ICU discharge, or death or a maximum of 30 days of follow-up)
  Incidence of delirium will be verified by trained intensive care professionals with the confusion assessment method for the ICU 2 times per day.

SECONDARY OUTCOMES:
Daily hazard of delirium among ICU patients | During ICU stay (from enrollment until ICU discharge, or death or a maximum of 30 days of follow-up)
  The daily hazard of delirium will be analyzed using a joint survival model that accounts for the treatment effect on repeated daily indicator of delirium (Confusion Assessment Method for the ICU) within each patient and terminating event (death or discharge from the ICU).
Antipsychotic use among ICU patients | During ICU stay (from enrollment until ICU discharge, or death or a maximum of 30 days of follow-up)
  Need of antipsychotic use during ICU stay
Need of mechanical restraints among ICU patients | During ICU stay (from randomization until ICU discharge, or death, or a maximum of 30 days of follow-up)
  Need of mechanical restraints among ICU patients during ICU stay
Coma-free days at day 7 among ICU patients | During the first 7 days following patient enrollment.
  Days alive and free of coma (Richmond Agitation Sedation Scale -4 or -5) during ICU stay.
Unplanned loss of invasive devices among ICU patients | During ICU stay (from randomization until ICU discharge, or death, or a maximum of 30 days of follow-up)
  Unplanned loss of venous catheter, tube feeding or urinary catheter
Mechanical ventilation-free days at day 7 among ICU patients | During the first 7 days following patient enrollment.
  Days alive and free of mechanical ventilation during ICU stay.
Any ICU-acquired infection among ICU patients | During ICU stay (from enrollment until ICU discharge, or death or a maximum of 30 days of follow-up)
  Pneumonia or bloodstream infection or urinary tract infection acquired after 48 hours of ICU admission.
ICU-acquired pneumonia among ICU patients | During ICU stay (from enrollment until ICU discharge, or death or a maximum of 30 days of follow-up)
  Pneumonia acquired after 48 hours of ICU admission.
ICU-acquired bloodstream infection among ICU patients | During ICU stay (from enrollment until ICU discharge, or death or a maximum of 30 days of follow-up)
  Bloodstream infection acquired after 48 hours of ICU admission.
ICU-acquired urinary tract infection among ICU patients | During ICU stay (from enrollment until ICU discharge, or death or a maximum of 30 days of follow-up)
  Urinary tract infection acquired after 48 hours of ICU admission.
ICU length of stay among ICU patients | During ICU stay (from enrollment until ICU discharge, or death or a maximum of 30 days of follow-up)
  Length of ICU stay in days
All-cause hospital mortality among ICU patients | During hospital stay (from enrollment until hospital discharge, or death or a maximum of 30 days of follow-up)
  rates of all-cause mortality during hospital stay
Symptoms of anxiety among family members | IOn the day of patient discharge from ICU, or death or a maximum of 30 days of follow-up.
  symptoms of anxiety among family members measured by the Hospital Anxiety and Depression scale
Symptoms of depression among family members | On the day of patient discharge from ICU, or death or a maximum of 30 days of follow-up.
  symptoms of depression among family members measured by the Hospital Anxiety and Depression scale
Satisfaction among among family members | On the day of patient discharge from ICU, or death or a maximum of 30 days of follow-up.
  Rates of patient's families satisfaction measured by the critical care family needs inventory
Prevalence of Burnout Syndrome among ICU professionals | It will be measured in two moments: within 15 days prior to the first ICU intervention and between the 15th and 30th days of the period in which no patient will be enrolled.
  Prevalence of Burnout Syndrome among ICU workers measured by the Maslach Burnout Inventory
Satisfaction with the current ICU visiting policy among ICU professionals | It will be measured between the 15th and 30th days of the period in which no patient will be enrolled.
  Satisfaction with the current ICU visiting policy among ICU professionals
Any adverse event related to ICU visitation | During ICU stay (from randomization until ICU discharge, or death, or a maximum of 30 days of follow-up)
  Any adverse event possible related to the ICU visitation model

CONTACTS AND LOCATIONS:
Overall Officials: Regis Rosa, MD, PhD, Principal Investigator — Hospital Moinhos de Vento
Locations (33):
- Brazil (33):
  - Hospital de Urgência e Emergência de Rio Branco, Rio Branco, Acre
  - Fundação Hospital Adriano Jorge, Manaus, Amazonas
  - Hospital Geral Clériston Andrade, Feira de Santana, Estado de Bahia
  - Hospital INCARDIO, Feira de Santana, Estado de Bahia
  - Hospital de Urgências de Goiânia, Goiânia, Goiás
  - Hospital das Clínicas da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Santa Casa de Misericórdia de São João Del Rei, São João del Rei, Minas Gerais
  - Hospital do Caâncer de Cascavel (UOPECCAN), Cascavel, Paraná
  - Hospital Universitário do Oeste do Paraná (UNIOESTE), Cascavel, Paraná
  - Hospital Universitário Alcides Carneiro, Campina Grande, Paraíba
  - Hospital Universitário Lauro Wanderley, João Pessoa, Paraíba
  - Hospital Regional do Baixo Amazonas, Santarém, Pará
  - Hospital Universitário de Petrolina, Petrolina, Pernambuco
  - Hospital Agamenom Magalhães, Recife, Pernambuco
  - Hospital Universitário da Universidade Federal do Piauí, Teresina, Piauí
  - Hospital Geral de Nova Iguaçú, Nova Iguaçu, Rio de Janeiro
  - Hospital Deoclécio Marques de Lucena, Parnamirim, Rio Grande do Norte
  - Hospital Tacchini, Bento Gonçalves, Rio Grande do Sul
  - Hospital São Camilo de Esteio, Esteio, Rio Grande do Sul
  - Hospital da Cidade de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Dom Vicente Scherer, Porto Alegre, Rio Grande do Sul
  - Hospital Mãe de Deus, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceiçaão, Porto Alegre, Rio Grande do Sul
  - Hospital Santa Rita, Porto Alegre, Rio Grande do Sul
  - Pavilhão Pereira Filho, Porto Alegre, Rio Grande do Sul
  - Hospital Ana Nery, Santa Cruz do Sul, Rio Grande do Sul
  - Hospital Santa Cruz, Santa Cruz do Sul, Rio Grande do Sul
  - Hospital Dona Helena, Joinville, Santa Catarina
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto, São Paulo
  - Hospital do Coração (HCor), São Paulo, São Paulo
  - Hospital Alberto Urquiza Wanderley (UNIMED João Pessoa), João Monlevade
  - Hospital Montenegro, Montenegro

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Rosa RG, Falavigna M, Robinson CC, da Silva DB, Kochhann R, de Moura RM, Santos MMS, Sganzerla D, Giordani NE, Eugenio C, Ribeiro T, Cavalcanti AB, Bozza F, Azevedo LCP, Machado FR, Salluh JIF, Pellegrini JAS, Moraes RB, Hochegger T, Amaral A, Teles JMM, da Luz LG, Barbosa MG, Birriel DC, Ferraz IL, Nobre V, Valentim HM, Correa E Castro L, Duarte PAD, Tregnago R, Barilli SLS, Brandao N, Giannini A, Teixeira C; ICU Visits Study Group Investigators and the BRICNet. Study protocol to assess the effectiveness and safety of a flexible family visitation model for delirium prevention in adult intensive care units: a cluster-randomised, crossover trial (The ICU Visits Study). BMJ Open. 2018 Apr 13;8(4):e021193. doi: 10.1136/bmjopen-2017-021193. PMID 29654049
- [Background] Sganzerla D, Teixeira C, Robinson CC, Kochhann R, Santos MMS, de Moura RM, Barbosa MG, da Silva DB, Ribeiro T, Eugenio C, Schneider D, Mariani D, Jeffman RW, Bozza F, Cavalcanti AB, Azevedo LCP, Machado FR, Salluh JI, Pellegrini JAS, Moraes RB, Damiani LP, da Silva NB, Falavigna M, Rosa RG. Statistical analysis plan for a cluster-randomized crossover trial comparing the effectiveness and safety of a flexible family visitation model for delirium prevention in adult intensive care units (the ICU Visits Study). Trials. 2018 Nov 19;19(1):636. doi: 10.1186/s13063-018-3006-8. PMID 30454019
- [Derived] de Souza JMB, Miozzo AP, da Rosa Minho Dos Santos R, Mocellin D, Rech GS, Trott G, Estivalete GPM, Sganzerla D, de Souza D, Rosa RG, Teixeira C. Long-term effects of flexible visitation in the intensive care unit on family members' mental health: 12-month results from a randomized clinical trial. Intensive Care Med. 2024 Oct;50(10):1614-1621. doi: 10.1007/s00134-024-07577-3. Epub 2024 Aug 22. PMID 39172240
- [Derived] Rosa RG, Pellegrini JAS, Moraes RB, Prieb RGG, Sganzerla D, Schneider D, Robinson CC, Kochhann R, da Silva DB, Amaral A, Prestes RM, Medeiros GS, Falavigna M, Teixeira C. Mechanism of a Flexible ICU Visiting Policy for Anxiety Symptoms Among Family Members in Brazil: A Path Mediation Analysis in a Cluster-Randomized Clinical Trial. Crit Care Med. 2021 Sep 1;49(9):1504-1512. doi: 10.1097/CCM.0000000000005037. PMID 33870915
- [Derived] Rosa RG, Falavigna M, da Silva DB, Sganzerla D, Santos MMS, Kochhann R, de Moura RM, Eugenio CS, Haack TDSR, Barbosa MG, Robinson CC, Schneider D, de Oliveira DM, Jeffman RW, Cavalcanti AB, Machado FR, Azevedo LCP, Salluh JIF, Pellegrini JAS, Moraes RB, Foernges RB, Torelly AP, Ayres LO, Duarte PAD, Lovato WJ, Sampaio PHS, de Oliveira Junior LC, Paranhos JLDR, Dantas ADS, de Brito PIPGG, Paulo EAP, Gallindo MAC, Pilau J, Valentim HM, Meira Teles JM, Nobre V, Birriel DC, Correa E Castro L, Specht AM, Medeiros GS, Tonietto TF, Mesquita EC, da Silva NB, Korte JE, Hammes LS, Giannini A, Bozza FA, Teixeira C; ICU Visits Study Group Investigators and the Brazilian Research in Intensive Care Network (BRICNet). Effect of Flexible Family Visitation on Delirium Among Patients in the Intensive Care Unit: The ICU Visits Randomized Clinical Trial. JAMA. 2019 Jul 16;322(3):216-228. doi: 10.1001/jama.2019.8766. PMID 31310297